CLINICAL TRIAL: NCT03895138
Title: A Feasibility Randomized Control Trial to Investigate the in Silico Optimization of Insulin Treatments
Brief Title: Trial to Investigate the in Silico Optimization of Insulin Treatments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Principal Investigator, Anthony McCall, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20164; 5R21EB018052 (NIH)
Record Dates: First submitted 2019-02-21; First posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-02

CONDITIONS: Coronary Artery Bypass

STUDY DESIGN:
Intervention Model Description: Subjects with CABG or open heart valve surgery will be enrolled in the study. They will be randomized to receive one of the following treatments:
  1. Standard Glucommander Protocol (SGP)
  2. Optimized Glucommander (OGM)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Glucommander Protocol (SGP) (Active Comparator): CABG or open valve surgery patients treated for stress hyperglycemia with the standard Glucomander protocol according to the manufacturer recommendations
  Interventions: Other: Standard Glucommander Protocol (SGP)
- Optimized Glucommander (OGM) (Experimental): CABG or open valve surgery patients treated for stress hyperglycemia with in silico optimized Glucomander protocol
  Interventions: Other: Optimized Glucommander (OGM)

INTERVENTIONS:
Other: Standard Glucommander Protocol (SGP) — Subjects receive standard Glucommander-based insulin therapy from the clinical staff of U.Va.'s cardiothoracic ICU and follow manufacturer's guidelines for starting with an initial multiplier value of .05.
  Arms: Standard Glucommander Protocol (SGP)
Other: Optimized Glucommander (OGM) — The experimental arm of the study involves treating subjects with a lower initial multiplier (.02 versus .05), a higher set of BG thresholds (140-180 mg/dl vs 120-160) in the first eight (8) hours of care for avoidance of hypoglycemia in that time period, and a requirement for consistent hourly-or-faster sampling of BG (as opposed to the Glucommander recommendation which is dependent on the trajectory of BG and can sometimes allow intervals of two hours between samples). After the eight (8) hours, the Glucommander is set back to the standard protocol for the entire duration of the subject's post-operative hospital stay.
  Arms: Optimized Glucommander (OGM)

SUMMARY:
The primary objective of this study is to assess the performance of an in silico designed alternative protocol for control of stress hyperglycemia of inpatients treated for Coronary Artery Bypass Graft (CABG) or valve replacement surgery in the University of Virginia cardiothoracic ICU.

DETAILED DESCRIPTION:
The hypothesis of the study is that settings for the Glucommander protocol can be optimized in silico to achieve statistically improved low blood glucose index (LBGI) within the subpopulation of CABG and valve replacement patients who both receive Glucommander-based insulin therapy and meet Manufacturer's guidelines for starting with an initial multiplier value of .052, without risking clinically significant increase in exposure to hyperglycemia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted for CABG and/or open heart valve surgery
2. Must have a 0.05 initial multiplier setting for the Glucommander based on the manufacturers recommendations
3. Age of 40-75, inclusive

Exclusion Criteria:

1. History of severe hypoglycemia within six months of hospital admission
2. Currently undergoing dialysis or renal replacement therapy
3. Women of childbearing potential
4. Patients with endocarditis needing valve replacement
5. Participation in another clinical trial at the time of screening.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2018-03-19 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Exposure to risk of hypoglycemia | 24 hours of post-operative hospital stay
  Exposure to risk of hypoglycemia as measured by the Low Blood Glucose Index (LBGI).

SECONDARY OUTCOMES:
Exposure to risk of hypoglycemia | 48 hours of post-operative hospital stay
  Exposure to risk of hypoglycemia as measured by the Low Blood Glucose Index (LBGI).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vrginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided